CLINICAL TRIAL: NCT07106775
Title: Evaluation of the Family Intervention Program (PIF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Gobierno de Cantabria (Unknown); Loyola University (Other); University of Jaen (Unknown)
Responsible Party: Principal Investigator, Victoria Hidalgo García, Principal Investigator, University of Seville
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRJ202304792
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Parenting; Children/Adolescent Adjustment; Family Functioning
Keywords: Positive parenting; Parenting competences; Program evaluation; Family functioning; Parenting practices; Effectiveness; Home program

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to the manualized program according to the inclusion criteria. The comparison group will be composed of families in areas where the intervention is not available but with similar sociodemographic characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Families receiving intervention (Experimental): Families who are participating in the home program
  Interventions: Behavioral: Family Intervention Program (PIF)
- Control group (No Intervention): Families who are not participating in the program and live in a comparable area where any of the intervention is offered

INTERVENTIONS:
Behavioral: Family Intervention Program (PIF) — Home psychoeducational intervention in an individual format driven by a practitioner where caregivers learn parenting competences and children learn autonomy and emotional regulation skills
  Arms: Families receiving intervention

SUMMARY:
The goal of this study is to evaluate the effectiveness of home positive parenting programs targeted to families at psychosocial risk carried out in Cantabria (Spain).

The investigators will collect information before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years). Besides, the investigators will compare these results with information from other families that are not taking part in the program. Depending on the case, the practitioners in charge of the intervention, the main caregivers of the participating families and/or the adolescents will provide the information for the study.

The investigators expect that families participating in the programs will improve their parenting competencies, their family dynamics, and the life quality of their children.

DETAILED DESCRIPTION:
A quasi-experimental design will be followed, with at least three evaluation moments and with a non-randomized comparison group.

Families will be referred to the PIF from social services. The participants will answer a series of questionnaires and scales, where they will give information related to sociodemographic data, parenting competencies, family functioning and children/adolescent adjustment. The information will be digitized through a computer application to which only the professional intervening with the family will have access. The app will not allow the participants to leave any question with no answer or with an incorrect answer.

To analyze the data, the investigators will use the softwares Mplus and Statistical Package for the Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Being a psychosocial at-risk family with at least one child under 18 years of age
* Living in the territory that corresponds to that social services center

Exclusion Criteria:

* Experience family crisis that prevent for participating in the home intervention
* Experience mental health issue that prevent for participating in the home intervention
* High level of psychosolcial risk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Family functioning | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  SCORE rated on a 5-point Likert-type scale ranging from 1 to 5. Higher scores mean a better outcome.
Children's quality of life | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  KIDSCREEN-10 rated on a 5-point Likert-type scale ranging from 1 to 5. Higher scores mean a better outcome.
Satisfaction with Family Life | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  Satisfaction with Family Life Scale (SWFLS), rated on a 7-point Likert-type scale ranging from 1 to 7. Higher scores mean a better outcome.
Emotional intelligence | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  The Emotional Quotient Inventory: Youth Version (EQ-i:YV) rated on a 4-point Likert-type scale ranging from 1 to 4. Higher scores mean a better outcome.
Indicators of social integration of the family | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  This ad hoc instrument rated on a 4-point Likert-type scale ranging from 1 to 4. Higher scores mean a better outcome.
Children adjustment | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  The Strengths and Difficulties Questionnaire (SDQ) rated on a 3-point Likert-type scale ranging from 0 to 2. Higher scores mean a better outcome.
School adjustment indicators | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  This ad hoc instrument rated on a 4-point Likert-type scale ranging from 1 to 4. Higher scores mean a better outcome.
Parental Competencies | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  The Parenting Competencies Assessment Interview (ECP - 12) rated on a 5-point Likert-type scale ranging from 1 to 5. Higher scores mean a better outcome.
Autonomy and life skills | Before the intervention, and every six months until the family achieves the proposed objectives (with a maximum intervention period of two years)
  The Life Skills Inventory (LSI) rated on a 2-point Likert-type scale ranging from 0 to 1. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Expectations about the intervention | Before the intervention
  This ad hoc instrument rated on a 4-point Likert-type scale ranging from 1 to 4. Higher scores mean a better outcome.
Perceived change after the intervention | Every six months from the start of the intervention until the family achieves the proposed objectives (with a maximum intervention period of two years)
  This ad hoc instrument rated on a 4-point Likert-type scale ranging from 1 to 4. Higher scores mean a better outcome.
Satisfaction with the intervention | Every six months from the start of the intervention until the family achieves the proposed objectives (with a maximum intervention period of two years)
  Client Satisfaction Questionnaire (CSQ-8), rated on a 4-point Likert-type scale ranging from 1 to 4. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Consejería de Inclusión Social, Juventud, Familias E Igualdad, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No
The project is framed in an agreement with the Govern of Cantabria and the researchers have no authorization for sharing individual participant data.

REFERENCES:
- [Background] Ugarriza Chávez, N., y Pajares Del Águila, L. (2005). La evaluación de la inteligencia emocional a través del inventario de BarOn ICE: NA, en una muestra de niños y adolescentes. Persona, 8, 11-58. https://www.redalyc.org/articulo.oa?id=147112816001
- [Background] Bar-On, R. (1997a). Development of the Baron EQ-I: A measure of emotional and social intelligence. 105th Annual Convention of the American Psychological Association in Chicago.
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Zabriskie, R. y McCormick, B. (2003). Parent and child perspectives of family leisure involvement and satisfaction with family life. Journal of Leisure Research, 35, 163-189. doi: 10.1080/00222216.2003.11949989
- [Background] Stratton, P., Bland, J., Janes, E. y Lask, J. (2010). Developing a practicable outcome measure for systemic family therapy: The SCORE. Journal of Family Therapy, 32, 232-258. doi: 10.1111/j.1467-6427.2010.00507.x
- [Background] European Kidscreen Groupe (2006). The KIDSCREEN questionnaires. Quality of life questionnaires for children and adolescents. Pabst Science Publ.
- See also: Report on the actions carried out for the advice and evaluation of the actions of the education and family intervention programs and services of the public social services of Cantabria — https://www.serviciossocialescantabria.org/uploads/documentos%20e%20informes/Evaluaci%C3%B3n%20Programas%20y%20Servicios%20de%20Educaci%C3%B3n%20e%20Intervenci%C3%B3n%20Familiar.pdf
- See also: Family Intervention Program (PIF): Technical manual for its implementation and evaluation — https://idus.us.es/items/566e83e8-e080-45e7-9356-3271cc52cafd